CLINICAL TRIAL: NCT05168254
Title: Clinical and Multiomics Study of First-line Chemotherapy for Advanced Pancreatic Cancer：a Prospective Single-center Research Trial
Brief Title: Clinical and Multiomics Study of First-line Chemotherapy for Advanced Pancreatic Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, duowu zou, Chief physician, Ruijin Hospital
Other Study IDs: RuijinH20201123
Record Dates: First submitted 2021-11-13; First posted 2021-12-23 (Actual); Last update posted 2021-12-23 (Actual); Status verified 2021-12

CONDITIONS: Pancreatic Ductal Adenocarcinoma, PDAC
MeSH Terms: conditions — Anophthalmia with pulmonary hypoplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — in situ tissue samples of pancreatic cancer by EUS-FNAare immediately sent to the laboratory for sequencing.
  Serum, plasma and peripheral blood mononuclear cells (PBMC) are isolated from peripheral blood samples; Serum and plasma are stored in - 80 ℃ refrigerator, and PBMC are stored in liquid nitrogen.
  Biological samples of all patients are kept in a regulated biological sample bank.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The early symptoms of pancreatic cancer are not obvious, and the early diagnosis rate is low. For most patients with pancreatic cancer,palliative chemotherapy is the only choice .At present, The guidance of NCCN guidelines on the selection of chemotherapy regimens for patients with advanced pancreatic cancer is only based on the physical condition(the ECOG score), which is one of the important reasons for the poor efficacy of chemotherapy in patients with advanced pancreatic cancer.Therefore, it is urgent to group pancreatic cancer patients according to tumor molecular typing and heterogeneity of response to chemotherapy drugs accurately,so as to guide the personalized treatment of patients.

DETAILED DESCRIPTION:
Based on the limitations of existing studies and the needs of clinical patients, the investigators chose two time points: after the diagnosis of pancreatic cancer (before the first-line chemotherapy), and after chemotherapy evaluation in this study, to obtain in situ samples of pancreatic cancer tissues by EUS-FNA.The samples are detected by dynamic multi-omics study before and after treatment(including genomics, transcriptomics, proteomics, metagenomics, etc.).Combined with the drug reaction and clinical outcome of patients, a comprehensive model is established to predict the clinical outcome of patients with PDAC and the choice of chemotherapy regimens, so as to screen the pancreatic cancer patients who are most likely to benefit from different chemotherapy regimens, and lay the foundation for the development of individual chemotherapy for advanced pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years old, male or female;
2. Locally advanced or metastatic pancreatic ductal adenocarcinoma confirmed by histopathology / cytology of the primary and / or metastatic lesions and not suitable for surgical resection, and don't receive chemotherapy;
3. According to the evaluation criteria of solid tumor efficacy(RECIST 1.1), there should be at least one measurable lesion (non nodular lesion with the longest diameter of 210 mm, or nodular lesion with the shortest diameter of more than 15 mm);
4. Patients voluntarily participate in this study, sign informed consent, have good compliance, and cooperate with follow-up.

Exclusion Criteria:

If any of the following criteria is met, the patient should be excluded:

1. Pancreatic ductal adenocarcinoma is diagnosed without histopathology / cytology;
2. The target lesion has received local non-drug therapy (including radiotherapy, physical and / or chemical ablation, etc.), and there is no imaging progression;
3. If the central nervous system metastasis is known, MRI should be performed to exclude it.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced pancreatic ductal adenocarcinoma
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of using the model to predict the therapeutic effect of drugs | 1.5 years
  The difference of progression free survival (PFS)

SECONDARY OUTCOMES:
Efficacy evaluation of solid tumor | 1.5 years
  disease control rate (DCR)
the quality of participants'life | 1.5 years
  According to the European Organization for research and treatment of cancer (EORTC) quality of life core scale EORTC QLQ-C30 (V3.0 Chinese version)，evaluating the quality of life (QOL)

CONTACTS AND LOCATIONS:
Overall Officials: Duowu Zou, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China